CLINICAL TRIAL: NCT06741410
Title: The Effect of Prophylactic Phenylephrine Infusion and Interventional Ephedrine Boluses on Umbilical Blood pH in Women Undergoing Cesarean Delivery Under Spinal Anesthesia: a Retrospective Case - Control Study
Brief Title: Ephedrine Versus Phenylephrine for Spinal Block - Related Hypotension in Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Bartosz Horosz, MD, Principal Investigator, Centre of Postgraduate Medical Education
Other Study IDs: 96/2024
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Spinal Anesthesia; Cesarean Delivery; Neonatal Acidosis
Keywords: cesarean delivery; spinal anesthesia; phenylephrine; ephedrine; hypotension
MeSH Terms: conditions — Hypotension | interventions — Ephedrine; Phenylephrine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ephedrine: Cesarean delivery cases where spinal block was administered and hypotension was managed with intravenous ephedrine.
  Hospital electronic database will be searched to identify cases of cesarean delivery in years 2020 - 2022. After that, manual review of the medical notes will follow in order to extract cases where spinal block was administered and ephedrine was used to treat spinal - related hypotension. Further chart analysis will yield demographic and hemodynamic data of the parturient, as well as clinical data of the neonate (weight, gender, Apgar score).
  Further laboratory data on neonatal acid - base status will be acquired from hospital's laboratory electronic database. Attention will be paid to assure that identification of the patients would not be possible using data acquired for the study. All data will be anonymized and accessible only for investigators.
  Interventions: Drug: Ephedrine
- Phenylephrine: Cesarean delivery cases where spinal block was administered and hypotension was managed with intravenous phenylephrine infusion
  Hospital electronic database will be searched to identify cases of cesarean delivery in years 2020 - 2022. After that, manual review of the medical notes will follow in order to extract cases where spinal block was administered and infusion of phenylephrine was used to treat spinal - related hypotension. Further chart analysis will yield demographic and hemodynamic data of the parturient, as well as clinical data of the neonate (weight, gender, Apgar score).
  Further laboratory data on neonatal acid - base status will be acquired from hospital's laboratory electronic database. Attention will be paid to assure that identification of the patients would not be possible using data acquired for the study. All data will be anonymized and accessible only for investigators.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Ephedrine — Intravenous boluses of ephedrine
  Groups: Ephedrine
Drug: Phenylephrine — Intravenous continuous infusion of phenylephrine
  Groups: Phenylephrine

SUMMARY:
The study is designed to compare two strategies used in the management of hypotension caused by spinal anesthesia for cesarean section: intravenous phenylephrine given as prophylactic infusion and interventional boluses of intravenous ephedrine. Phenylephrine is currently recommended for battling spinal anesthesia - related sympathectomy, due to some scientific data on possible negative effects of ephedrine on fetal wellbeing. Therefore this study will retrospectively compare both clinical and laboratory data of the newborns delivered by cesarean section where either large dose of ephedrine or continuous infusion of phenylephrine was used for management of hypotension

DETAILED DESCRIPTION:
Single - shot spinal block is a gold standard of anesthesia for cesarean delivery. It has been proven to decrease maternal morbidity and improve neonatal outcomes. Despite being most frequently used type of anesthesia in obstetrics, spinal block - related complications remain frequent in term parturients, of which hypotension is of utmost importance. Two widely accepted medications used in its prevention and treatment are phenylephrine and ephedrine, of which continuous, preventive phenylephrine infusion is considered superior in terms of neonatal safety.

Although there is some scientific evidence towards ephedrine having negative effect on neonatal acid - base status, it is still the most popular vasoconstrictor used for management of perioperative hypotension in Poland. It is an indirect adrenergic agonist, acting through release of noradrenaline from peripheral nerve endings. Beta - receptors mediated adrenergic stimulation of neonatal tissues is thought to be responsible for endocrine abnormalities, acid - base disturbances and possibly worse Apgar scores. Phenylephrine on the other hand is a direct and selective alpha-1 agonist and is regarded to exert very little or even no neonatal effects. Maternal complications related to phenylephrine infusion is hypertension and reflex bradycardia.

As convincing evidence is still lacking, this study is designed to retrospectively compare neonatal outcomes and perioperative hemodynamic data of mothers where either infusion of phenylephrine or boluses of ephedrine were used to control spinal -related hypotension during cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery at term under spinal anesthesia
* American Society of Anesthesiologists (ASA) physical status <3
* BMI <40
* Preemptive phenylephrine infusion or ephedrine boluses used during surgical procedure

Exclusion Criteria:

* No vasoconstrictor (phenylephrine nor ephedrine) used throughout the procedure
* Total dose of ephedrine less than 15mg
* poor quality of anesthetic record - data required for analysis not available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initial cohort of patients will consist of selected cases of cesarean deliveries from Orlowski Hospital in years 2020 - 2022, Department of Obstetrics and Gynaecology, Warsaw, Poland.
  Intention is to include 40 cases in each group.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Umbilical blood pH | During delivery (from spinal injection to umbilical clamping and cutting)
  Sets of data will be tested for normality and standard statistical tests (Student's t - test or Mann - Whitney U - test) will be used to detect the differences in umbilical blood pH between the groups.
Umbilical blood Base Excess (BE) | During delivery (from spinal injection to umbilical clamping and cutting)
  Sets of data will be tested for normality and standard statistical tests (Student's t - test or Mann - Whitney U - test) will be used to detect the differences in umbilical blood Base Excess (BE) between the groups.

SECONDARY OUTCOMES:
Hemodynamic stability | During delivery (from spinal injection to umbilical clamping and cutting)
  Number of episodes of hypotension recorded in anesthetic sheet after spinal injection will be compared using chi-square or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Malec-Milewska, MD, Prof., Study Chair — Department of Anesthesia and Intensive Care, Orlowski Hospital, Warsaw
Locations (1):
- Centre of Postgraduate Medical Education,Department of Anesthesia and Intensive Care, Warsaw, Poland

REFERENCES:
- [Background] Ngan Kee WD, Khaw KS, Tan PE, Ng FF, Karmakar MK. Placental transfer and fetal metabolic effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology. 2009 Sep;111(3):506-12. doi: 10.1097/ALN.0b013e3181b160a3. PMID 19672175
- [Background] Higgins N, Fitzgerald PC, van Dyk D, Dyer RA, Rodriguez N, McCarthy RJ, Wong CA. The Effect of Prophylactic Phenylephrine and Ephedrine Infusions on Umbilical Artery Blood pH in Women With Preeclampsia Undergoing Cesarean Delivery With Spinal Anesthesia: A Randomized, Double-Blind Trial. Anesth Analg. 2018 Jun;126(6):1999-2006. doi: 10.1213/ANE.0000000000002524. PMID 28953494
- [Background] Mohta M, Aggarwal M, Sethi AK, Harisinghani P, Guleria K. Randomized double-blind comparison of ephedrine and phenylephrine for management of post-spinal hypotension in potential fetal compromise. Int J Obstet Anesth. 2016 Aug;27:32-40. doi: 10.1016/j.ijoa.2016.02.004. Epub 2016 Feb 21. PMID 27020488